CLINICAL TRIAL: NCT05496036
Title: Neoadjuvant PD-1 Blockade in Resectable Merkel Cell Carcinoma
Acronym: MCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 01622
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab (Experimental): Study participants will undergo a tumor tissue collection biopsy prior to treatment, followed by one dose of pembrolizumab 400mg, then undergo a curative intent resection of all remaining disease 3 weeks after the initial dose of pembrolizumab. Post-operatively, subjects will receive up to 1 year of pembrolizumab 400mg every 6 weeks.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 400mg IV
  Other Names: Keytruda

SUMMARY:
The main purpose of this study is to determine the response of Merkel cell carcinoma to pembrolizumab before surgery and to determine whether it further reduces the risk for disease recurrence. Another purpose of this study is to look at the side effects that occur when the experimental drug pembrolizumab is given to people with Merkel cell carcinoma before and after their standard of care surgery to remove the Merkel cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Must have resectable stage I-III MCC.
2. Must be expected to have an adequate amount of tumor burden to yield 2-4 pre-operative research core biopsy (14-gauge needle) specimens or the equivalent amount of tissue (4-6 mm punch biopsy), in addition, to the tissue required for diagnostic purposes. For stage III MCC patients, assessment of measurable disease/tumor burden will be determined by tumor imaging and reviewed by the treatment team.
3. Must be expected to have an adequate amount of residual tumor after their pre-operative research tumor tissue collection, such that their operative research tumor collection will also yield at least 4-6 research core biopsy specimens or the equivalent amount of tissue.
4. Must be willing to undergo the two paired tumor tissue biopsy procedures to obtain samples for biomarker analysis. Tissue obtained must not be previously irradiated.
5. Male subjects must agree to use a contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
6. Female subjects must not be pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) OR a WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
7. Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
9. Have adequate organ function.
10. Hepatitis B (HBV) positive subjects

    * Subjects who is HBsAg positive is eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.
    * Subject should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.
11. Subject with history of Hepatitis C (HCV) infection are eligible if HCV viral load is undetectable at screening. Subject must have completed curative anti-viral therapy at least 4 weeks prior to randomization.

Exclusion Criteria:

1. Have unresectable disease; i.e. in the opinion of the surgical oncologist, all of the subject's MCC cannot be completely removed with a clear margin.
2. If the subject had major surgery, the subject must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention
3. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation.
4. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
5. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.
6. Has received prior radiotherapy within 2 weeks of start of study intervention. Subject must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
7. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
8. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
9. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
10. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Subject with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
11. Has known active CNS metastases and/or carcinomatous meningitis. Subject with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
12. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
14. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
15. Has an active infection requiring systemic therapy.
16. Has a known history of Human Immunodeficiency Virus (HIV) infection.
17. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
21. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
: Pathologic Response Rate | Approximately 3 weeks
  The number of subjects with pathologic complete response (CR) or near CR defined by less than 10% viable tumor cells will be determined for subjects who received 1 dose of neoadjuvant pembrolizumab and underwent definitive surgery. PathCR/nearCR rate is defined as the percentage of treated subjects who achieve PathCR/nearCR

SECONDARY OUTCOMES:
Frequency and incidence of adverse events | Up to 13 months
  Toxicity will be determined by scoring treatment-related AEs and SAEs. CTCAE version 5.0 grades will be employed.
Tumor infiltrating response (TIL) | Approximately 3 weeks
  Patients will be assessed for TIL response at the 3-week resection time point, with the resection tumor assessed for tumor-infiltrating lymphocytes by a board-certified pathologist. TIL response will be captured as a binary outcome that is either brisk TIL (diffuse lymphocytes throughout the tumor) or not (non-brisk TIL or absent TIL)
Two Year Recurrence-Free Survival | Approximately 2 years
  Recurrence-free survival (RFS) is defined as the time from date of surgery to date of disease recurrence, death due to any cause or most recent follow-up documenting freedom from recurrence (i.e., scan date).

CONTACTS AND LOCATIONS:
Overall Officials: John Miura, MD, Principal Investigator — Penn Medicine
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No